CLINICAL TRIAL: NCT05454072
Title: SinoNasal Microbiota Transfer (SNMT) to Treat Chronic Rhinosinusitis: A Randomized, Double-blind, Placebo-controlled Trial
Brief Title: Microbiota Transfer for Chronic Rhinosinusitis
Acronym: SNMT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Amin Javer (Other)
Responsible Party: Sponsor-Investigator, Amin Javer, Clinical Professor, St. Paul's Hospital, Canada
Organization: St. Paul's Hospital, Canada (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H18-02263-A013
Record Dates: First submitted 2022-07-07; First posted 2022-07-12 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: Sinusitis, Chronic; Sinus Disease; Sinus Infection; Sinus Infection Chronic
Keywords: Microbiota Transplant; Chronic Rhinosinusitis
MeSH Terms: conditions — Sinusitis; Bronchiolitis Obliterans Syndrome; Paranasal Sinus Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sinonasal Microbiota Transfer (Experimental): The transfer site for patients will be prepared by endoscopically removing any visible crusting, mucin, and purulent discharge from the sinuses and via manual high-volume (>60 ml), high-pressure saline wash on day 0. The donor mucus sample will be homogenized using sterile, disposable rotor-stator homogenizer tips for 30 seconds and 5 ml of donor mucus will be instilled into the affected sinus cavity(ies) using a masked syringe under endoscopic visualization, with the recipient's head in a dependent position. Patients will remain in this position for 15 minutes to facilitate transfer.
  Interventions: Procedure: Sinonasal Microbiota Transfer
- Sham Sinonasal Microbiota Transfer (Sham Comparator): Sterile saline will replace the SNMT donor mucus in the masked syringe and will be delivered in an identical manner to the SNMT intervention.
  Interventions: Procedure: Sham Sinonasal Microbiota Transfer

INTERVENTIONS:
Procedure: Sinonasal Microbiota Transfer — Pre-screened donor mucus, up to 15mL, will be transplanted into each diseased sinus via nasal lavage.
  Arms: Sinonasal Microbiota Transfer
Procedure: Sham Sinonasal Microbiota Transfer — Saline, up to 15mL, will be transplanted into each diseased sinus via nasal lavage.
  Arms: Sham Sinonasal Microbiota Transfer

SUMMARY:
Chronic sinusitis (CRS) is a common inflammatory condition of the sinuses that affects up to 2.5% of the Canadian population, and is thought to be caused by bacterial infection, resistant biofilms, chronic inflammation and possibly an unhealthy population of sinus microbes (or microbiota). Symptoms include nasal obstruction and discharge, facial pain, loss of smell and sleep disturbance, which all strongly impact quality of life. CRS treatment involves nasal or oral steroids, repeated rounds of antibiotic, and sinus surgery. Despite maximal treatment, some recalcitrant patients suffer with CRS for years.

The lack of new, effective therapies to treat CRS leads the investigators to test whether a SinoNasal Microbiota Transfer (SNMT) could trigger CRS recovery. SNMT is defined as the endoscopic transfer of a healthy sinus microbiota from a fully screened donor's sinus to a CRS patient's sinus(es). Similar to a fecal transplant used to treat Clostridioides difficile diarrhea, the sinonasal microbiota transfer may eliminate sinus pathogens and restore the sinus microbiota to a healthy state. SNMT will be combined with a one-time, high volume, high pressure "sinus power wash" pre-treatment to temporarily clear the way for the donor microbiota to establish itself. The investigators will conduct a proof-of-principle, randomized, double-blind, placebo-controlled trial of 80 subjects to test whether a sinus power wash plus SNMT improves clinical outcomes in CRS patients.

DETAILED DESCRIPTION:
Chronic rhinosinusitis (CRS) is a common inflammatory condition of the paranasal sinuses. CRS patients experience persistent facial pain/pressure, nasal discharge, nasal obstruction, and loss of smell. Initial treatment includes topical and systemic steroids and (often multiple rounds of) antibiotics; however, two thirds of patients remain symptomatic despite medical therapy and require endoscopic sinus surgery. Direct medical and indirect social costs of CRS are substantial, with 57% of patients reporting absenteeism and poor health and 28% experiencing associated anxiety and depression. These hard-to-treat patients are classified as recalcitrant CRS (rCRS), have limited treatment options available, and are the focus of this trial.

CRS was thought to occur due to impaired sinus ventilation and drainage however new evidence suggests that sinus mucosal inflammation, driven in part by microbiota disruptions and pathogen carriage, is the etiological factor behind CRS. Type of inflammation varies and cannot be predicted based on clinical variables alone. Several studies show that the microbiome composition of CRS patients is less diverse compared to healthy subjects, suggesting that community-level disruptions, and not individual opportunistic pathogens, may contribute to persistent inflammation.

The investigators will conduct a proof-of-principle, randomized, double-blind, placebo-controlled trial of 80 subjects to test whether a sinus power wash plus SNMT improves clinical outcomes in CRS patients within 45 days compared to a sinus power wash and sham SNMT. The investigators will investigate the safety profile of SNMT and determine if SNMT-related CRS symptom improvement lasts up to 6 months. Finally, the investigators will investigate how SNMT contributes to CRS recovery, by tracking changes in the sinus microbiota and inflammation pre- and post-treatment. Results from our pilot study shows that SNMT produced CRS symptom improvement in 75% of patients. SNMT therapy may be a transformative strategy to address CRS, a chronic and debilitating illness.

ELIGIBILITY:
Inclusion Criteria for Patients:

* Recalcitrant CRS patients
* Able to provide informed consent
* Diagnosed with CRS (with/without polyps) and have previously undergone functional endoscopic sinus surgery (Post-FESS)
* Continued to fail despite receiving "maximal and adequate medical treatment" This is defined as patients who:
* Have received topical nasal steroids in any form (Spray/ Rinse/ Atomized) for at least 3 months or at least one course of oral corticosteroids treatment (>0.5 mg/kg for 2 weeks tapering dose);
* Had at least one course of antibiotic treatment either based on culture and sensitivity of nasal sinus secretions or as long-term low dose macrolide therapy (clarithromycin 500mg twice a day for 2 weeks then 250 mg once a day for 4 weeks) for at least one trial or have received a course of itraconazole 100mg twice daily for 6 weeks
* Have deteriorating SNOT-22 Scores (≥20) or do not improve after surgery and appropriate maximal medical management (MLK score ≥ 2, with at least 2 points on the discharge subdomain)

Exclusion Criteria for Patients:

* Diagnosed with sinonasal tumors
* Autoimmune diseases affecting the upper airway (e.g., systemic lupus erythematosus, Sjögren's syndrome, systemic sclerosis)
* Immune-compromised patients
* Impairment in mucociliary function (e.g., cystic fibrosis, Kartagener syndrome)
* Pregnant or planning to become pregnant or breastfeeding
* Severe underlying disease with anticipated survival less than 6 months
* Unable to tolerate SNMT for any reason

Inclusion Criteria for Donors:

* 19 years of age or older
* Able to provide informed consent, complete donor screening, and adhere to SNMT mucus collection and testing procedures

Exclusion Criteria for Donors:

* If they are positive for any of the following: (i) from blood or mucus testing, human Immunodeficiency virus (HIV) I/II, hepatitis A IgM, hepatitis B surface antigen (HBsAg), hepatitis C, human T- lymphotropic virus (HTLV) I/II, methicillin-resistant Staphylococcus aureus, multidrug resistant bacteria, and/or SARS-CoV-2
* A history of sinonasal or lower airway disease within the last 2 years other than the common cold; diagnosed with CRS; diagnosed with acute rhinosinusitis within the last six months; asthma; and/or clinical findings of sinonasal disease at the inclusion visit and immunodeficiency; any history of active cancer, or risk factors for acquisition of HIV, syphilis, hepatitis A, hepatitis B, hepatitis C, prion, or relevant neurological disease, receipt of blood transfusion from a country other than Canada in the preceding 6 months, any type of antibiotic treatment or any systemic immunosuppressive agents in the 3 months prior to the donation, or any current or previous medical or psychosocial condition or behaviours, which in the opinion of the investigator, may pose a risk to the recipient or the donor

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-06-15 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Modified Lund-Kennedy (MLK) endoscopic scoring | Baseline to 45 days
  Change in endoscopic score, where points to each sinus are assigned based on discharge (0 - no discharge; 1 - clear discharge; 2 - purulent discharge), edema (0 - edema; 1 - mild edema; 2 - severe edema), and polyps (0 - no polyps; 1 - confined to the middle meatus; 2 - beyond the middle meatus) for a maximum of 6 points per side (12 total). A 1-point difference in the total MLK score is considered clinically meaningful since it signifies a change in either polyp size, edema severity, or type of discharge.

SECONDARY OUTCOMES:
Sinonasal Outcome Test (SNOT-22) questionnaire | Baseline to 45 days, 90 days, 180 days
  Disease specific quality of life improvement, which includes 22 questions that encompass 4 subdomains of CRS (nasal, sleep, otologic/facial pain, and emotional symptoms).
Smell Test | Baseline to 45 days, 90 days, 180 days
  Smell test using Sniffin' Sticks (scores range from 0-48).
Adverse and serious adverse events | Baseline to any time until the end of the study period
  The safety of SNMT will be examined by identifying any adverse events, including serious adverse events.
Microbiome analysis of patients and donor samples | Baseline to 45 days, 90 days, 180 days
  Metagenome sequencing will be performed to construct metagenome-assembled genomes of CRS pathogens in donor and recipient mucus, to unambiguously describe strain-specific eradication or reinfection; determine donor sinus microbiota engraftment; detect evidence for (or not) resistance gene and resistant organism transfer via SNMT from donor to recipient; and investigate microbiome compositional and functional features associated with SNMT success or failure.
Immune markers | Baseline to 45 days, 90 days, 180 days
  To assess immune activation and inflammation-related responses to SNMT CRS-specific structured histological analysis will be performed to detect a reduction in tissue eosinophilia and/or neutrophilia, mucosal ulceration, and squamous metaplasia; cytokine/chemokine testing to detect a decrease in inflammation; and antibody testing and blood work to measure sustained reductions in serum eosinophils and IgE levels

CONTACTS AND LOCATIONS:
Overall Officials: Amin Javer, MD, Study Director — University of British Columbia
Locations (1):
- St. Paul's Hospital, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lange B, Holst R, Thilsing T, Baelum J, Kjeldsen A. Quality of life and associated factors in persons with chronic rhinosinusitis in the general population: a prospective questionnaire and clinical cross-sectional study. Clin Otolaryngol. 2013 Dec;38(6):474-80. doi: 10.1111/coa.12189. PMID 24131818
- [Background] Smith KA, Orlandi RR, Rudmik L. Cost of adult chronic rhinosinusitis: A systematic review. Laryngoscope. 2015 Jul;125(7):1547-56. doi: 10.1002/lary.25180. Epub 2015 Jan 30. PMID 25640115
- [Background] Macdonald KI, McNally JD, Massoud E. The health and resource utilization of Canadians with chronic rhinosinusitis. Laryngoscope. 2009 Jan;119(1):184-9. doi: 10.1002/lary.20034. PMID 19117310
- [Background] Baguley C, Brownlow A, Yeung K, Pratt E, Sacks R, Harvey R. The fate of chronic rhinosinusitis sufferers after maximal medical therapy. Int Forum Allergy Rhinol. 2014 Jul;4(7):525-32. doi: 10.1002/alr.21315. Epub 2014 Mar 7. PMID 24610673
- [Background] Stein NR, Jafari A, DeConde AS. Revision rates and time to revision following endoscopic sinus surgery: A large database analysis. Laryngoscope. 2018 Jan;128(1):31-36. doi: 10.1002/lary.26741. Epub 2017 Jul 8. PMID 28688189